CLINICAL TRIAL: NCT01966796
Title: Clinical Characteristics and Microbiology of Healthcare Associated Pneumonia
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ping-Huai Wang, Medical Dr, Far Eastern Memorial Hospital
Other Study IDs: 102013-E
Record Dates: First submitted 2013-10-12; First posted 2013-10-22 (Estimated); Results first posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Healthcare Associated Pneumonia
Keywords: healthcare associated pneumonia; drug-resistant bacteria; pneumonia severity index
MeSH Terms: conditions — Healthcare-Associated Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- PSI II: PSI less than 70 or equal to 70
- PSI III: PSI 70-90
- PSI IV: PSI 90-130
- PSI V: PSI more than 130

SUMMARY:
Background The prediction of multi-drug resistant (MDR) pathogens is a key issue in the management of health-care associated pneumonia (HCAP). Multiple risk factors have been proposed, some of which overlap with items of the pneumonia severity index (PSI). The aim of this study was to investigate the relationship between PSI and presence of MDR pathogens.

Methods Patients who were admitted to a tertiary-care hospital from January 2005 to December 2010 were screened by a discharge diagnosis of pneumonia. Patients were enrolled if they fulfilled the definition of HCAP by 2005 ATS/IDSA guideline.

DETAILED DESCRIPTION:
MDR bacteria were defined as Pseudomonas aeruginosa (P. aeruginosa), Enterobacter species, those not sensitive to second and third generation cephalosporins, Acinetobacter species, extended-spectrum β-lactamase (ESBL) Enterobacteriaceae such as Escherichia coli (E. coli) and Klebsiella pneumoniae (K. pneumoniae), Burkholderia cepacia (B. cepacia), Stenotrophomonas maltophilia (S. maltophilia), and methicillin resistant Staphylococcus aureus (MRSA).

The criteria for HCAP is defined as follows: patients who had been hospitalized in an acute care hospital for two or more days within the past 90 days; residents of a nursing home or long-term care facility; recipients of recent intravenous antibiotic therapy, chemotherapy or wound care within the past 30 days; or patients who attended a hospital or hemodialysis clinic.

ELIGIBILITY:
Inclusion Criteria:

* patients who had been hospitalized in an acute care hospital for two or more days within the past 90 days;
* residents of a nursing home or long-term care facility;
* recipients of recent intravenous antibiotic therapy, chemotherapy or wound care within the past 30 days;
* or patients who attended a hospital or hemodialysis clinic.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were admitted to the Far Eastern Memorial Hospital, an 800-bed tertiary care hospital in northern Taiwan, from January 2005 to December 2010 were screened by discharge diagnoses.The patients whose primary discharge diagnosis was pneumonia (International Classification of Diseases codes 482, 485, and 486) were selected.
Sampling Method: Probability Sample
Enrollment: 530 (Actual)
Dates: Start 2013-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ping-huai Wang, M.D., Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

REFERENCES:
- [Background] Bartlett JG, Dowell SF, Mandell LA, File TM Jr, Musher DM, Fine MJ. Practice guidelines for the management of community-acquired pneumonia in adults. Infectious Diseases Society of America. Clin Infect Dis. 2000 Aug;31(2):347-82. doi: 10.1086/313954. Epub 2000 Sep 7. No abstract available. PMID 10987697
- [Background] Hospital-acquired pneumonia in adults: diagnosis, assessment of severity, initial antimicrobial therapy, and preventive strategies. A consensus statement, American Thoracic Society, November 1995. Am J Respir Crit Care Med. 1996 May;153(5):1711-25. doi: 10.1164/ajrccm.153.5.8630626. No abstract available.
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Background] Micek ST, Reichley RM, Kollef MH. Health care-associated pneumonia (HCAP): empiric antibiotics targeting methicillin-resistant Staphylococcus aureus (MRSA) and Pseudomonas aeruginosa predict optimal outcome. Medicine (Baltimore). 2011 Nov;90(6):390-395. doi: 10.1097/MD.0b013e318239cf0a. PMID 22033455
- [Background] Song JH, Oh WS, Kang CI, Chung DR, Peck KR, Ko KS, Yeom JS, Kim CK, Kim SW, Chang HH, Kim YS, Jung SI, Tong Z, Wang Q, Huang SG, Liu JW, Lalitha MK, Tan BH, Van PH, Carlos CC, So T; Asian Network for Surveillance of Resistant Pathogens Study Group. Epidemiology and clinical outcomes of community-acquired pneumonia in adult patients in Asian countries: a prospective study by the Asian network for surveillance of resistant pathogens. Int J Antimicrob Agents. 2008 Feb;31(2):107-14. doi: 10.1016/j.ijantimicag.2007.09.014. Epub 2007 Dec 26. PMID 18162378

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who were admitted to our hospital,Jan 2005 to Dec 2010 The patients with the diagnosis was pneumonia were selected. They were enrolled if they fulfilled the criteria for HCAP defined in 2005 ATS/IDSA
Groups:
- PSI II: Pneumonia severity index less than 70 or equal to 70, (Pneumonia is more severe if the index is higher)
- PSI III: Pneumonia severity index 70-90
- PSI IV: Pneumonia severity index 91-130
- PSI V: Pneumonia severity index more than 130
Period: Overall Study
Arm/Group | PSI II | PSI III | PSI IV | PSI V
Started | 15 | 51 | 195 | 269
Completed | 15 | 51 | 195 | 269
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PSI II | PSI III | PSI IV | PSI V | Total
Number analyzed (Participants) | 15 | 51 | 195 | 269 | 530
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 21 | 50 | 17 | 100
  >=65 years | 3 | 30 | 145 | 252 | 430
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (12.5) | 66.4 (11.7) | 73.3 (12.5) | 79.5 (10.2) | 75.1 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 20 | 56 | 100 | 181
  Male | 10 | 31 | 139 | 169 | 349
Region of Enrollment [Number; unit: participants]
  Taiwan | 15 | 51 | 195 | 269 | 530

OUTCOME MEASURES:

1. Primary Outcome: Pathogens of Healthcare Associated Pneumonia, Measured by the Number of Participants
Description: sputum culture and sterile specimen such as blood or pleural effusion culture for healthcare associated pneumonia within seven days of admission
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | PSI II | PSI III | PSI IV | PSI V
Number analyzed (Participants) | 15 | 51 | 195 | 269
Participants | 15 | 51 | 195 | 269

2. Primary Outcome: Number of Participants With MDR Pathogens
Description: MDR bacteria were defined as Pseudomonas aeruginosa (P. aeruginosa), Enterobacter species, those not sensitive to second and third generation cephalosporins, Acinetobacter species, extended-spectrum β-lactamase (ESBL) Enterobacteriaceae such as Escherichia coli (E. coli) and Klebsiella pneumoniae (K. pneumoniae), Burkholderia cepacia (B. cepacia), Stenotrophomonas maltophilia (S. maltophilia), and methicillin resistant Staphylococcus aureus (MRSA).
Time Frame: seven days after admission
Measure: Number; unit: participants
Arm/Group | PSI II | PSI III | PSI IV | PSI V
Number analyzed (Participants) | 15 | 51 | 195 | 269
participants
  MDR | 1 | 13 | 72 | 120
  mortality | 0 | 3 | 24 | 64
Statistical Analysis 1: Comparison: PSI II vs PSI III vs PSI IV vs PSI V; The incidence of MDR pathogens (6.7%, 25.5%, 36.9% and 44.6% in PSI II, III, IV, and V, respectively, p=0.002) and mortality rate (0, 5.9%, 12.3%, and 23.8%, respectively, p<0.001) increased with increasing PSI; Test type: Superiority or Other; p = 0.002, ANOVA

ADVERSE EVENTS:
Description: It was a retrospective observational study. No intervention was done during this study. Thereafter, no serious adverse event was assessed.
Arm/Group | PSI II | PSI III | PSI IV | PSI V
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PSI II (N=0) | PSI III (N=0) | PSI IV (N=0) | PSI V (N=0)
Serious adverse event (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — It was a retrospective observational study. No intervention was done during this study. Thereafter, no serious adverse event was assessed.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PSI II (N=0) | PSI III (N=0) | PSI IV (N=0) | PSI V (N=0)
non-serious adverse event (Investigations) | 0 | 0 | 0 | 0 — It was a retrospective observational study. No intervention was done during this study. Thereafter, no adverse event was assessed.

LIMITATIONS AND CAVEATS:
The limitations to this study is that the microbiology data mainly came from sputum cultures, retrospective studies and single center experience

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No